CLINICAL TRIAL: NCT04794244
Title: Healthy Living in Overweight and Obese Adolescents ASGE-FABES Program in Development of Formats Effect:Randomized Controlled Study
Brief Title: Healthy Living in Overweight and Obese Adolescents ASGE-FABES Program in Development of Formats
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: aysun ardıç (Other)
Responsible Party: Sponsor-Investigator, aysun ardıç, Ph.D. lecturer, lead researcher, Istanbul University - Cerrahpasa
Organization: Istanbul University - Cerrahpasa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Project number: 116S210; 116S210 (Other Grant/Funding Number: The Scientific and Technological Research Council of Turkey)
Record Dates: First submitted 2021-03-02; First posted 2021-03-12 (Actual); Last update posted 2021-03-12 (Actual); Status verified 2021-03

CONDITIONS: Healthy Lifestyle Behaviors; Overweight Adolescents; Obese Adolescents
Keywords: Adolescent health; nursing; obesity; school health; healthy lifestyle behaviors
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): group in which the experimental group training program is applied
  Interventions: Behavioral: ASGE-FABES Program
- No Intervention (No Intervention): group without control group training program

INTERVENTIONS:
Behavioral: ASGE-FABES Program — In the control group study, pretest-posttest and experimental design with repeated measurements were used in randomized groups. An overweight and obese adolescent constituted the sample of 250 (125-experiment, 125-control) of the study. Research data Socio-Demographic Features Information Form, Adolescent Nutrition Information Scale, Adolescent Physical Activity Information Scale, Adolescent Lifestyle Scale, Healthy Lifestyle Choice Scale for Adolescents, Beck Anxiety Scale, Daily Food Consumption Form, Beverage Consumption Form, collected using. Data are saved before and after application. ASGEFABES PROGRAM was applied to the experimental group for 10 weeks. Measurements after the training program were collected in four measurements: 1st week, 6th and 12th months.
  Arms: Experimental

SUMMARY:
The aim of this project is to develop multiple behavioral strategies for the prevention of obesity in adolescents.

ASGE-FABES [Adolescent Health Promotion Physical Activity, Physical activity of overweight and obese youth of Nutrition, Stress Management] Program,to evaluate its effects on nutrition and mental health. Program overweight and obeseadolescents to lose weight in a healthy way, healthy lifestyle behaviors make healthy choices, nutritional and physical activity knowledgecognitive and It aims to gain behavioral skills. In the study, "pretest-posttest in randomized groupswith control group, with repeated measures & quot; experimental design type is used. The sample of the research,250 (125-experiment, 125-control) constituted an overweight and obese adolescent.

DETAILED DESCRIPTION:
The aim of this project is to evaluate the impact of ASGE-FABES Program for the prevention of obesity in adolescents on physical activity, nutritional and mental health of overweight and obese adolescents. The program aims at promoting cognitive and behavioral skills for overweight and obese adolescents to lose weight in a healthy way, to promote healthy lifestyle behaviors, to make healthy choices, to increase their knowledge of nutrition and physical activity, to assume their own health responsibilities and to cope with stress. In the study, quot;experimental design type with randomized groups, pretest-posttest control group, repeated measurement" was used. The sample of the study consisted of 250 overweight and obese adolescents studying in the 6th grade of 10 secondary schools in Şişli district of Istanbul. The data of the study were collected using with Socio-Demographic Characteristics Form,Adolescent Nutrition Information Scale,Adolescent Physical Activity Information Scale, Adolescent Lifestyle Scale, Adolescent Healthy Lifestyle Choose Scale, Beck Anxiety Scale, Daily Food Consumption Form and Beverage Consumption Form.The data were collected before the application, at the first week after the application, and at the sixth and 12th months. Descriptive statistical tests, pearson chi-square tests, t-test in similar groups, repeated measures anova, and Cohen's effect size tests were used in the analysis of the study. There was no significant difference between the experimental and control groups in terms of the descriptive characteristics, behavioral and cognitive variables of adolescents.

ELIGIBILITY:
Inclusion Criteria:

* being overweight or obese
* 11-12 age range
* children asked by their parents to participate in the study

Exclusion Criteria:

* having a genetic disease
* normal weight
* mental disability

Ages: 11 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Actual)
Dates: Start 2017-09-20 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2019-07-09 (Actual)

PRIMARY OUTCOMES:
body measurements | "through study completion, an average of 1 year".
  The results of this study are the results of the ASGE-FABES program. In this study, body measurements include calculating body mass index. BKI is calculated as kg / m ^ 2.

CONTACTS AND LOCATIONS:
Overall Officials: aysun ARDIÇ, Ph.D, Principal Investigator — Istanbul University - Cerrahpasa
Locations (1):
- İstanbul University-Cerrahpaşa, Istanbul, İ̇stanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I reserve the data sharing as it is promised to the subjects that the data sharing will be kept confidential.